CLINICAL TRIAL: NCT02941029
Title: RADTOX: Measuring Radiation Toxicity Using Circulating DNA
Acronym: RADTOX
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: DiaCarta, Inc. (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201601961-N; 261201600063C-0-0-1 (NIH); OCR15535 (Other: OnCore)
Record Dates: First submitted 2016-10-13; First posted 2016-10-21 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer
Keywords: Radiation; Chemotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — collection of plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Evaluate toxicity biomarkers: Investigators will determine if measurement of circulating DNA from tumor and normal tissues shortly after RT provides an early and quantitative measure of risk of radiation-related complications. It will be necessary to collect blood specimens prior to and during the first week of radiation therapy.
  Interventions: Other: Plasma Blood collection

INTERVENTIONS:
Other: Plasma Blood collection — Plasma blood collection is collected at specific intervals prior to and during radiation treatment.
  Other Names: Plasma/Blood Collection

SUMMARY:
This research study is being done to develop a new test to identify prostate cancer patients at highest risk of radiotherapy-related complications. This research study would allow monitoring of total tissue damage within 24 hours of radiation exposure in blood samples that could give an initial result within a few days that would help clinicians make treatment decisions. Detection of unusual tissue damage at this early time, well before symptoms occur, could allow doctors to tailor interventions that could include patient therapies that would reduce or prevent the problems that occur due to treatment of their cancer.

DETAILED DESCRIPTION:
Currently, a patient's risk for toxicity is based almost exclusively on population statistics. Radiation (and chemotherapy) dose are based on phase I data and not on the individual's specific genetics or hidden predispositions. RadTox measures cell damage within 24 hours of radiation exposure and should help identify patients at higher risk for radiation complications. This should allow physicians to adjust radiation field size and dose to minimize long-term toxicity.

Patients undergoing radiation treatment for stage I to III prostate cancer, using protons or X-rays, either as primary treatment or consolidation after prostatectomy (positive margins or prostate-specific assay [PSA]-related indications) will be eligible. Hormone treatment will be allowed.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in the study and a signed and dated an institutional review board (IRB)-approved consent form conforming to federal and institutional guidelines.
* ≥ 18 years of age.
* Patients must have an Eastern Cooperative Oncology Group (An ECOG) performance status of 0 or 1.
* A diagnosis of adenocarcinoma of the prostate.
* Not yet begun definitive therapy with chemotherapy or radiation but may have hormones or surgery.
* Clinically stage I to III tumors.

Exclusion Criteria:

* Metastatic disease.
* A history of invasive rectal malignancy or other pelvic malignancy, regardless of disease-free interval.
* Active inflammatory bowel disease (i.e., patients requiring current medical interventions or who are symptomatic).
* Prior pelvic radiation therapy for any reason.
* Psychiatric or addictive disorders or other conditions that, in the opinion of the principal investigator (PI), would preclude the patient from meeting the study requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients with undergoing radiation therapy for prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Free circulating DNA will be measured in patients undergoing radiation for prostate cancer as a toxicity biomarker compared to CTCAE v4.0 | 9 Months

SECONDARY OUTCOMES:
Free circulating DNA will be measured in patients undergoing radiation for prostate cancer as a toxicity biomarker compared pain scores | 9 Months
Free circulating DNA will be measured in patients undergoing radiation for prostate cancer as a toxicity biomarker compared and visual analog scales of toxicity | 9 Months

CONTACTS AND LOCATIONS:
Overall Officials: Randal Henderson, MD, MBA, Principal Investigator — clinical professor
Locations (2):
- United States (2):
  - University of Florida Health, Gainesville, Florida
  - University of Florida Health Proton Therapy Institute, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No
Data will be shared with necessary government agencies, the sponsor, and participating providers and institutions as defined in the informed consent document.